CLINICAL TRIAL: NCT07036250
Title: A Single-arm, Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of U32 Injection in Patients With Acute Myeloid Leukemia.
Brief Title: Clinical Study of U32 in Patients With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U32-03
Record Dates: First submitted 2025-05-27; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukaemia
Keywords: CAR-T; CD38; CLL-1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- U32 CAR-T cells (Experimental): The Patients will be enrolled into 3 dose level cohorts
  Interventions: Drug: U32 CAR-T

INTERVENTIONS:
Drug: U32 CAR-T — Lymphodepletion preconditioning is required prior to CAR-T cell therapy. Lymphodepletion will be performed using a regimen of cyclophosphamide (250-500 mg/m²) and fludarabine (25-30 mg/m²), each administered for 3 consecutive days.

SUMMARY:
This is a single-arm, open-label clinical study to evaluate the safety, tolerability, and efficacy of U32 injection in patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of U32 in the treatment of acute myeloid leukemia and to determine the safe and effective dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and be expected to complete the follow-up examinations and treatments as required by the study protocol.
2. Be aged ≥2 years and ≤65 years at the time of signing the informed consent form, with no restrictions on gender.
3. Meet the AML diagnosis according to the 2022 WHO classification and satisfy the diagnostic criteria for relapsed and refractory acute myeloid leukemia as defined in the "Chinese Guidelines for the Diagnosis and Treatment of Relapsed and Refractory Acute Myeloid Leukemia (2023 Edition)": a) Relapsed AML diagnostic criteria: reappearance of leukemia cells in peripheral blood after complete remission (CR), or positivity for minimal residual disease (MRD) detected by flow cytometry in bone marrow (excluding other causes such as bone marrow regeneration after consolidation chemotherapy), or extramedullary infiltration of leukemia cells. b) Refractory AML diagnostic criteria: newly diagnosed cases that are ineffective after two courses of standard treatment; relapse within 12 months after CR and subsequent consolidation therapy; relapse after 12 months that is ineffective to conventional chemotherapy; cases with two or more relapses; persistent extramedullary leukemia.
4. AML patients who are molecularly positive after treatment and cannot achieve negativity through conventional therapy.
5. Positive expression of CD38 or CLL-1 confirmed by immunohistochemistry or flow cytometry.
6. Have previously received at least two lines of adequate treatment or allogeneic hematopoietic stem cell transplantation (HSCT).
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 3, with an expected survival of more than 3 months.
8. Have adequate bone marrow reserve at screening, defined as: absolute lymphocyte count (ALC) ≥0.3×10^9/L, platelets (PLT) ≥20×10^9/L (including with platelet transfusion support).
9. Have appropriate organ function: aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN); alanine aminotransferase (ALT) ≤3 times ULN; total bilirubin ≤1.5 times ULN; serum creatinine ≤1.5 times ULN, or creatinine clearance rate ≥60 mL/min; hemoglobin ≥60 g/L or maintained at this level after transfusion; peripheral capillary oxygen saturation ≥92%; left ventricular ejection fraction (LVEF) ≥45%.
10. Female subjects must meet the following criteria to be considered for enrollment: a) Be of non-childbearing potential, defined as: having undergone hysterectomy or bilateral oophorectomy, or having had bilateral tubal ligation, or being postmenopausal (complete cessation of menstruation for ≥1 year); b) Be of childbearing potential, but have a negative serum pregnancy test at screening, and agree to use medically accepted contraceptive measures (such as intrauterine device, oral contraceptives, or condoms) before enrollment and during the study, until 1 year after the last study drug administration.
11. Male subjects of childbearing potential must agree to use barrier contraception or complete abstinence until 1 year after the last study drug administration.
12. Have sufficient venous access for apheresis or intravenous blood draw, and no contraindications for leukapheresis.
13. For subjects who have received daratumumab or other CD38 - targeted therapies, the washout period for CD38 monoclonal antibody should be at least 3 months before the reinfusion treatment.

Exclusion Criteria:

1. Having other malignancies within 3 years prior to screening, with the exception of adequately treated cervical carcinoma in situ, papillary thyroid carcinoma, basal cell carcinoma or squamous cell carcinoma of the skin, localized prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery.
2. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), with detectable HBV-DNA levels above the lower limit of detection in peripheral blood; positive for hepatitis C virus (HCV) antibodies with detectable HCV-RNA levels above the lower limit of detection; positive for human immunodeficiency virus (HIV) antibodies; positive for cytomegalovirus (CMV) DNA; positive for EBV-DNA; positive for syphilis serology.
3. A history of severe allergic reactions [defined as allergic reactions of grade 2 or higher, with any of the following clinical manifestations: airway obstruction (rhinorrhea, cough, wheezing, dyspnea), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), urinary or fecal incontinence, laryngeal edema, bronchial spasm, cyanosis, shock, respiratory or cardiac arrest] or known allergy to any active ingredient, excipient, or murine product or xenoprotein contained in the study drug (including the lymphodepletion regimen).
4. Severe cardiac disease, including but not limited to severe arrhythmias, unstable angina, large myocardial infarction, New York Heart Association (NYHA) Class III or IV heart failure, refractory hypertension (defined as failure to achieve target blood pressure despite the use of a reasonable and tolerable regimen of ≥3 antihypertensive medications [including diuretics] for >1 month or requiring ≥4 antihypertensive medications for effective blood pressure control).
5. History of solid organ transplant or planned solid organ transplant (excluding allogeneic hematopoietic stem cell transplant).
6. Acute or chronic graft-versus-host disease (GVHD) that is deemed uncontrollable by the investigator.
7. Allogeneic hematopoietic stem cell transplant within 6 months prior to screening.
8. Active autoimmune or inflammatory disease (e.g., Guillain-Barré syndrome [GBS], amyotrophic lateral sclerosis [ALS]) or clinically significant active cerebrovascular disease (e.g., cerebral edema, posterior reversible encephalopathy syndrome [PRES]).
9. Presence of a tumor emergency (e.g., spinal cord compression, bowel obstruction, leukostasis, tumor lysis syndrome) requiring urgent treatment prior to screening or infusion.
10. Presence of uncontrollable bacterial, fungal, viral, or other infections requiring antibiotic therapy.
11. Planned to undergo major surgery within 4 weeks prior to lymphodepletion or during the study period, or surgical wounds not fully healed prior to enrollment.
12. Presence of severe psychiatric disorders.
13. Within 1 week prior to planned PBMC collection, receiving systemic corticosteroids or immunosuppressive agents that are deemed by the investigator to affect cell preparation. a) Systemic corticosteroids: subjects receiving systemic corticosteroid therapy within 1 week prior to planned PBMC collection and deemed by the investigator to require long-term systemic corticosteroid therapy during the treatment period (excluding inhaled or topical use); b) Immunosuppressive agents: subjects receiving immunosuppressive agents within 1 week prior to planned PBMC collection.
14. Received live-attenuated or live virus vaccines within 4 weeks prior to screening.
15. History of alcoholism or drug abuse.
16. Participation in another interventional clinical trial within 30 days prior to screening.
17. Any subject deemed by the investigator, based on clinical judgment or standards of care, to have a contraindication to any study procedure or other medical conditions that may pose an unacceptable risk.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after U32CAR-T cells infusion [Safety and Tolerability] | 28 days post administration of CAR-T-cells
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

SECONDARY OUTCOMES:
Pharmacokinetics of U32 CAR-T cells | 2 years post CAR T cell infusion
  Time at the maximal concentration(Tmax)
Pharmacokinetics of U32 CAR-T cells | 2 years post CAR T cell infusion
  Area under the concentration-time curve(AUC)
Pharmacokinetics of U32 CAR-T cells | 2 years post CAR T cell infusion
  The maximal concentration of eripheral blood (Cmax)
Pharmacodynamics of U32 CAR-T cells | 2 years post CAR T cell infusion
  Concentration levels of CAR-T-related serum cytokines such as IL-6, IFN γ, ferritin and CRP at each time point
Objective Response Rate (ORR), as assessed by Investigators | 2 years post CAR T cell infusion
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Remission (CR) or CR with partial hematologic recovery (CRh) or CR with incomplete hematologic recovery (CRi)
Duration of response (DOR), as assessed by Investigators | 2 years post CAR T cell infusion
  Duration of response (DOR) is defined as the time from the first documented objective response to the first documented disease progression or death.
Overall survival (OS) | 2 years post CAR T cell infusion
  Overall Survival (OS) was defined as the time from the date of first infusion of U32 to the date of death due to any cause.
Progression-free survival (PFS), as assessed by Investigators | 2 years post CAR T cell infusion
  Progression-free survival (PFS) was defined as the time from the date of infusion to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, JiangSu 215000 Recruiting, Suzhou, China